CLINICAL TRIAL: NCT03793530
Title: The Use of Bone Marrow Concentrate in Elective Tranforaminal Lumbar Interbody Fusion Surgery: A Randomized Control Trial
Brief Title: Autologous Bone Marrow Concentrate in Elective Tranforaminal Lumbar Interbody Fusion Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pei-Yuan Lee, MD (Other)
Collaborators: Aeon Biotechnology Corporation (Industry)
Responsible Party: Sponsor-Investigator, Pei-Yuan Lee, MD, Principal Investigator, Show Chwan Memorial Hospital
Organization: Show Chwan Memorial Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: RD106050
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Bone Marrow; Spinal Fusion
Keywords: Bone Marrow; Mesenchymal Stromal Cells; spine fusion surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bone marrow concentration group (Experimental): Transforaminal lumbar interbody fusion with local bone graft and intraoperative bone marrow concentration
  Interventions: Other: Transforaminal lumbar interbody fusion with local bone graft and intraoperative bone marrow concentration
- Control group (Active Comparator): Transforaminal lumbar interbody fusion with local bone graft
  Interventions: Other: Transforaminal lumbar interbody fusion with local bone graft

INTERVENTIONS:
Other: Transforaminal lumbar interbody fusion with local bone graft and intraoperative bone marrow concentration — Transforaminal lumbar interbody fusion with local bone graft and intraoperative bone marrow concentration
  Arms: Bone marrow concentration group
Other: Transforaminal lumbar interbody fusion with local bone graft — Transforaminal lumbar interbody fusion with local bone graft
  Arms: Control group

SUMMARY:
This study aims to evaluate the effect of bone marrow concentration on bone healing and spinal fusion by comparing clinical and imaging outcomes between patients receiving transforaminal lumbar intebody fusion with local bone graft and with intraoperative bone marrow concentration and those receiving transforaminal lumbar intebody fusion with local bone graft only.

DETAILED DESCRIPTION:
Spinal arthrodesis has become the mainstay of treatment for severe spinal deformity, spinal instability, spondylolisthesis, and symptomatic degenerative disease. Its primary goal is to develop an osseous bridge between adjacent motion segments to prevent motion, relieve pain, and facilitate neurological recovery. One of the arthrodesis method is transforaminal lumbar intebody fusion. After removal of the problematic disc, iliac crest bone graft was harvested and impacted into the space with cage to facilitate fusion. However, patients are exposed to additional risk of harvesting site, such as pain, infection, wound healing problem or hematomas. Local bone graft harvested from decompression is one of the alternative solutions to avoid these complications. However, the effect of local boen graft is inferior to iliac crest bone graft because iliac crest bone graft contains three important ingredients for successful fusion: osteoconductive scaffold, osteoinductive factors, and the ability to osteogenesis. Mesenchymal stem cells (MSCs) are pluripotent cells that can differentiate into multiple mesenchymal tissues, including tenocytes, chondrocytes and osteoblasts, as well as being a source of multiple growth factors to establish an environment conducive to soft and hard tissue regeneration. As bone marrow concentration has high concentration of mesenchymal stem cells, some studies have shown that autologous bone marrow concentration can improve bone healing. In this study, we will add bone marrow concentration into local bone graft during transforaminal lumbar intebody fusion and evaluate the effect of bone marrow concentration on bone healing and spinal fusion.

ELIGIBILITY:
Inclusion Criteria:

* With indication of transforaminal lumbar decomprassion and interbody fusion, ex. spondylolisthesis, symptomatic degenerative disease, spinal instability.
* Involved levels between T12 and S1
* Involved levels less than three levels
* Age between 20 and 70 years

Exclusion Criteria:

* With prior history of spinal surgery
* With current or prior history of tumor, trauma or infection at spine
* With current diagnosis of coagulopathy
* With current or prior history of cancer
* With current or prior history of hematological disease
* Pregnancy
* Patients who will not cooperate with one-year followup

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2017-08-01 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
3-month postoperative spinal function evaluated by Oswestry Disability Index | 3-month postoperative
  Subjective evaluation of spinal function by Oswestry Disability Index. Oswestry Disability Index ranges from 0 to 100 and lower score indicates less disability.

SECONDARY OUTCOMES:
6-month postoperative spinal function evaluated by Oswestry Disability Index | 6-month postoperative
  Subjective evaluation of spinal function by Oswestry Disability Index. Oswestry Disability Index ranges from 0 to 100 and lower score indicates less disability.
12-month postoperative spinal function evaluated by Oswestry Disability Index | 12-month postoperative
  Subjective evaluation of spinal function by Oswestry Disability Index. Oswestry Disability Index ranges from 0 to 100 and lower score indicates less disability.
3-month postoperative degree of pain evaluated by visual analogue scale | 3-month postoperative
  Subjective evaluation of degree of pain by visual analogue scale. Visual analogue scale for pain ranges from 0 to 10 and higher score indicates more pain.
6-month postoperative degree of pain evaluated by visual analogue scale | 6-month postoperative
  Subjective evaluation of degree of pain by visual analogue scale. Visual analogue scale for pain ranges from 0 to 10 and higher score indicates more pain.
12-month postoperative degree of pain evaluated by visual analogue scale | 12-month postoperative
  Subjective evaluation of degree of pain by visual analogue scale. Visual analogue scale for pain ranges from 0 to 10 and higher score indicates more pain.
3-month postoperative degree of bone healing evaluated by plain radiograph | 3-month postoperative
  Degree of bone healing evaluated by plain radiograph
6-month postoperative degree of bone healing evaluated by plain radiograph | 6-month postoperative
  Degree of bone healing evaluated by plain radiograph
12-month postoperative degree of bone healing evaluated by plain radiograph | 12-month postoperative
  Degree of bone healing evaluated by plain radiograph
12-month postoperative degree of bone healing evaluated by computed tomograph | 12-month postoperative
  Degree of bone healing evaluated by computed tomograph

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yuan Lee, MD, Study Chair — Show Chwan Memorial Hospital
Locations (1):
- Show Chwan Memorial Hospital, Changhua, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu MH, Tseng YK, Chung YH, Wu NY, Li CH, Lee PY. The efficacy of oral vitamin D supplements on fusion outcome in patients receiving elective lumbar spinal fusion-a randomized control trial. BMC Musculoskelet Disord. 2022 Nov 18;23(1):996. doi: 10.1186/s12891-022-05948-9. PMID 36401234